CLINICAL TRIAL: NCT00138021
Title: Cognitive Remediation in Supported Employment at HSC
Brief Title: Cognitive Remediation in Supported Employment at Human Service Center (HSC)
Acronym: CT+SE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Human Service Center, Illinois (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05 -132
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2007-11-02 (Estimated); Status verified 2007-10

CONDITIONS: Vocational Rehabilitation; Schizophrenia; Mental Disorders; Cognitive Symptoms
Keywords: Serious mental illness; Supported Employment; Cognitive remediation; Cognitive impairments
MeSH Terms: conditions — Schizophrenia; Mental Disorders; Neurobehavioral Manifestations; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Computerized cognitive training program — The cognitive training model used in the McGurk et al. (2005) study is referred to as the "Thinking Skills for Work" program. The program is a manualized, remediative and compensatory training intervention that is integrated with SE services. The program includes a cognitive trainer, a structured training manual (McGurk & Mueser, unpublished training manual) and a computer-based cognitive training program (described below).
  Other Names: The computerized cognitive training program using the Cogpack Software, version 7.4 (Marker Software, 2005).

SUMMARY:
This project seeks to evaluate the feasibility and effectiveness of combining cognitive remediation and Supported Employment Program (SEP) services to improve work outcomes in people with a serious mental illness who have been unable to benefit from vocational services (i.e., acquire or maintain a job). Cognitive remediation involves treating and improving cognitive impairments, such as memory (e.g., short-term and working memory), attention span, or problem solving skills. It is hypothesized that cognitive remediation will significantly improve peoples' employment outcomes in a supported employment program.

DETAILED DESCRIPTION:
Ample evidence documents that supported employment is an effective strategy for improving the vocational outcomes of persons with schizophrenia and other severe mental illnesses. However, a significant amount of clients receiving supported employment services work little or not at all. With respect to factors that may influence the work outcomes of persons participating in supported employment programs, cognitive functioning appears to be potentially important. Cognitive impairment in persons with severe mental illness (SMI) is strongly correlated with functional adjustment in the community and has been shown to be correlated with work, both contemporaneously and prospectively. Studies have demonstrated that clients who did not receive the full benefits of supported employment had more deficits in executive functioning, memory, and psychomotor speed than those clients who had better work outcomes.

The current study will use a computerized cognitive training program that will be administered by a cognitive trainer. The program consists of 24 training modules (each one takes about one hour to complete). Clients in an SEP who have been unable to maintain a job that they acquired while in the program can participate in the research. Clients who have agreed to participate in the research project will be randomly assigned to either receive the computerized training and supported employment services (CT-SES) or supported employment services (SES) without the training (i.e., treatment-as-usual-condition). Both research groups will receive the same baseline, three-month, and 12-month follow up interviews that will consists of a brief clinical and neuropsychological evaluation, an assessment of problems associated with finding or maintaining employment, and employment outcomes while enrolled in the study. In addition, both groups will receive a telephonic interview at 18 and 24 months to assess their employment outcomes (clinical and neurological information will not be collected at 18 or 24 months).

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in a Supported Employment Program
* Has acquired and lost at least one job while in the Supported Employment Program
* Presently unemployed

Exclusion Criteria:

* Has not acquired at least one job while in the Supported Employment Program
* Presently employed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-07; Study Completion 2008-05 (Estimated)

PRIMARY OUTCOMES:
competitive employment status at 12, 18, and 24 months | 12, 18, and 24 months
number of days employed in a competitive job at 12, 18, and 24 months | at 12, 18, and 24 months
number of jobs acquired and lost at 12, 18, and 24 months | at 12, 18, and 24 months

SECONDARY OUTCOMES:
improvement in cognitive functioning (various measures of cognitive functioning) at 3, 12, 18, and 24 months | 3, 12, 18, and 24 months
retention in either research condition | 3 & 12 months
clinical status at 3, 12, 18, and 24 months | 3, 12, 18, and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: David Loveland, Ph.D., Principal Investigator — Fayette Companies
Locations (1):
- Human Service Center (HSC), Peoria, Illinois, United States

REFERENCES:
- [Background] McGurk SR, Mueser KT, Pascaris A. Cognitive training and supported employment for persons with severe mental illness: one-year results from a randomized controlled trial. Schizophr Bull. 2005 Oct;31(4):898-909. doi: 10.1093/schbul/sbi037. Epub 2005 Aug 3. PMID 16079391